CLINICAL TRIAL: NCT05196724
Title: Holding a Foster Child's Mind in Mind
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: University of Copenhagen (Other); University College Copenhagen (Other); Anna Freud National Centre for Children and Families (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 301703
Record Dates: First submitted 2021-12-16; First posted 2022-01-19 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Attachment Disorder; Behavior Problem
Keywords: Foster care; Mentalization; Therapy; Attachment; Effects
MeSH Terms: conditions — Mental Disorders | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Intervention Model Description: This is a prospective cluster-randomized controlled trial with two conditions: (1) an intervention group who will receive MBT and (2) and a control group who receive usual care (UC).
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded for allocation when coding story stem and video outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentalization Based Therapy (MBT) (Experimental): MBT for foster carers is a 12 session therapeutic intervention that will be offered to foster families by municipal foster care consultants
  Interventions: Behavioral: Mentalization Based Therapy MBT
- Usual care (Active Comparator): the control group will receive the usual care offered to foster families such as supervision
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Mentalization Based Therapy MBT — The focus is on improving the core components of secure attachment, particularly by developing the reflective functioning for all professionals working with children in out-of-home care, which is subsequently proposed to increase the psychosocial adjustment of the child and decrease emotional and behavioral problems. MBT treatment consists of up to 12 weekly sessions with the foster parents and child covering three core components: 1) psycho-education about mentalizing, trauma, and attachment for foster parents; 2) support for reflective practice in the professional network, and 3) mentalization-based therapy for the foster family [41].
  Arms: Mentalization Based Therapy (MBT)
Behavioral: Usual care — The control group will receive the usual care offered to foster families such as supervision
  Arms: Usual care

SUMMARY:
The aim of this study is to examine the effects of Mentalization Based Therapy (MBT) for foster families in Denmark on child mental health and well-being, parental stress, mental health, and reflective function, parental mind-mindedness and the parent-child relationship.

DETAILED DESCRIPTION:
Children placed in foster care are psychologically and physically vulnerable and show more social, developmental, and behavioral problems than children living with their family of origin. Many foster parents struggle to care for these children, some of whom have experienced serious adversity at a young age. The study examines the effects of Mentalization Based Therapy (MBT) in a cluster-randomized controlled trial with 175 foster families with children aged 4-17 years in 10 Danish municipalities.

ELIGIBILITY:
Inclusion Criteria:

* Any kind of foster family (including professional and kinship care) with at least one full-time foster child aged 4-17 years.
* Elevated child symptoms as measured by X scales and
* An expressed need for support from either the foster parents or the foster child.

Exclusion Criteria:

* Foster families in which there are no reported difficulties and concerns regarding the child or the placement.
* Foster families in which the child was placed with the family within the last X months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Child mental health | post-intervention (16 weeks)
  The Child Behavior Checklist (CBCL) measures behavioral and emotional problems in children and adolescents. The CBCL consists of 113 questions, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). The CBCL is completed by foster parents for all children in the trial, and the Youth Self-Report (YSR) is completed by the foster children or adolescents aged 11 and above. The CBCL is widely used and has proven to be a useful tool for detecting psychopathology in children and shows good results regarding both validity and reliability

SECONDARY OUTCOMES:
Child Mental health | Follow-up (6 months post-intervention)
  The Child Behavior Checklist (CBCL) measures behavioral and emotional problems in children and adolescents. The CBCL consists of 113 questions, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). The CBCL is completed by foster parents for all children in the trial, and the Youth Self-Report (YSR) is completed by the foster children or adolescents aged 11 and above. The CBCL is widely used and has proven to be a useful tool for detecting psychopathology in children and shows good results regarding both validity and reliability
Child well-being | post-intervention (16 weeks)
  Kidscreen-10 is a 10-item measure of child well-being health-related quality of health). Items are scored from 1 (never) to 5 (always) except for items 1 and 9 (reverse). A higher score is better. Kidscreen-10 is used with families where the target foster child is 8 years old or more.
Child well-being | follow-up (6 months post-intervention)
  Kidscreen-10 is a 10-item measure of child well-being health-related quality of health). Items are scored from 1 (never) to 5 (always) except for items 1 and 9 (reverse). A higher score is better. Kidscreen-10 is used with families where the target foster child is 8 years old or more.
Parental reflective function | post-intervention (16 weeks)
  Parental Reflective Functioning Questionnaire - PRFQ is an 18 item measure of parental reflective function. The PRFQ consists of three subscales with score ranges 6-42: 1) Pre-Mentalizing Modes (PRFQ-PM) 6 items (a low score indicates better function). 2) Certainty about Mental States (PRFQ-CMS) 6 items (a medium score indicates better function). 3) Interest and curiosity in mental states PRFQ-IC 6 items (a high score indicates better function)
Parental reflective function | follow-up (6 months post-intervention)
  Parental Reflective Functioning Questionnaire - PRFQ is an 18 item measure of parental reflective function. The PRFQ consists of three subscales with score ranges 6-42: 1) Pre-Mentalizing Modes (PRFQ-PM) 6 items (a low score indicates better function). 2) Certainty about Mental States (PRFQ-CMS) 6 items (a medium score indicates better function). 3) Interest and curiosity in mental states PRFQ-IC 6 items (a high score indicates better function)
Parent-child interaction | post-intervention (16 weeks)
  To assess the foster parent-child relationship, the study uses the video-based system Coding Interactive Behavior (CIB). The CIB is a global rating system for social interactions that includes 22 parent codes, 16 child codes, and 5 dyadic codes rated on a scale of 1 to 5 which can be aggregated into the following composites: sensitivity, intrusiveness, limit setting, involvement, withdrawal, compliance, dyadic reciprocity, and dyadic negative states. The CIB is coded based on a 6-minute parent/child free-play or interaction recorded in the home or at another location if preferred by the family. The CIB system has been validated as an assessment measure in multiple studies of mother-child interactions in both normative and high-risk populations and shows stability over time, predictive validity, and adequate psychometric properties. The video will be with the child and one of the foster parents. The foster parents are free to choose which parent participates.
Attachment | post-intervention (16 weeks)
  The Story Stem Assessment Profile (SSAP) is a narrative-based measure, for the assessment of internal representations in children between the ages of 4 and 11 years old. Using a standard doll family and play materials, the interviewer enacts the beginning of a story (a story stem) and asks the child to complete the story using the provided play materials. The method allows the child to enact the story in a playful manner creating a narrative based on both verbal and nonverbal inputs, offering a unique insight into the child's perception of the nature and quality of relationships. The short version of the SSAP entails a set of 7 story stems, which introduce the beginning of a story for the child to complete, within which lies "an inherent dilemma." The SSAP has demonstrated robust psychometric properties and has been validated with children in out-of-home-care the UK.
Parental stress | post-intervention (16 weeks)
  The Parenting Stress Scale (PSS) [52,53] is an 18 item measure of parenting stress that is rated on a five-point scale (Strongly disagree, Disagree, Undecided, Agree, Strongly agree). Total score range 18-90, where a low score indicates less stress
Parental stress | follow-up (6 months post-intervention)
  The Parenting Stress Scale (PSS) [52,53] is an 18 item measure of parenting stress that is rated on a five-point scale (Strongly disagree, Disagree, Undecided, Agree, Strongly agree). Total score range 18-90, where a low score indicates less stress
Parent mental health | post-intervention (16 weeks)
  The WHO-5 index is a short questionnaire assessing emotional well-being in adults during the previous 2 weeks. It consists of five positively formulated items. The degree to which these feelings were present in the last 2 weeks is scored on a 6-point Likert-type scale ranging from 0 (not present) to 5 (constantly present). Item scores are summated and transformed to a 0-100 scale, with lower scores indicating poorer well-being. The WHO-5 index has been cross-culturally validated and has proven to be psychometrically sound.
Parent mental health | follow-up (6 months post-intervention)
  The WHO-5 index is a short questionnaire assessing emotional well-being in adults during the previous 2 weeks. It consists of five positively formulated items. The degree to which these feelings were present in the last 2 weeks is scored on a 6-point Likert-type scale ranging from 0 (not present) to 5 (constantly present). Item scores are summated and transformed to a 0-100 scale, with lower scores indicating poorer well-being. The WHO-5 index has been cross-culturally validated and has proven to be psychometrically sound.
Parental mind-mindedness | post-intervention (16 weeks)
  To assess representational Mind-mindedness we will use the mind-mindedness interview, addressing the foster carer's tendency to spontaneously think of the child as a psychological being. The foster carers will be asked to describe their child, and their answers are coded following the manual. The number of produced sentences about the child's mental characteristics (instead of sentences related to the child's behavior, physical or situational aspects) provides an indication of the level of the caregiver's mental representation of the child, or "representational mind-mindedness".
Parental mind-mindedness | follow-up (6 months post-intervention)
  To assess representational Mind-mindedness we will use the mind-mindedness interview, addressing the foster carer's tendency to spontaneously think of the child as a psychological being. The foster carers will be asked to describe their child, and their answers are coded following the manual. The number of produced sentences about the child's mental characteristics (instead of sentences related to the child's behavior, physical or situational aspects) provides an indication of the level of the caregiver's mental representation of the child, or "representational mind-mindedness".
Perception of the family | post-intervention (16 weeks)
  the general functioning subscale of the Family Assessment Device (FAD) is a 6-item subscale to measure the perception of the family function. It is scored on a 4-point Likert scale. Items are summed to a total subscale score
Perception of the family | follow-up (6 months post-intervention)
  the general functioning subscale of the Family Assessment Device (FAD) is a 6-item subscale to measure the perception of the family function. It is scored on a 4-point Likert scale. Items are summed to a total subscale score

CONTACTS AND LOCATIONS:
Overall Officials: Maiken Pontoppidan, PhD, Principal Investigator — VIVE
Locations (1):
- VIVE - The Danish Centre of Social Science Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the study are not publicly available to protect participant privacy but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Dalgaard NT, Villumsen AMA, Sorensen KM, Midgley N, Vaever MS, Almlund M, Pontoppidan M. Holding a foster child's mind in mind: study protocol for a cluster-randomized controlled trial of mentalization-based therapy (MBT) for foster families. BMC Psychol. 2023 Mar 7;11(1):62. doi: 10.1186/s40359-023-01103-8. PMID 36879301